CLINICAL TRIAL: NCT02300402
Title: Automatic Detection and Characterization of Residual Masses in Patients With Lymphomas Through Fusion of Whole-Body Diffusion-Weighted MRI on 3 Tesla and 18F-Fluorodeoxyglucose PET/CT
Brief Title: Detection and Characterization of Residual Masses in Lymphomas
Acronym: ADAMANTIUS
Status: Completed | Type: Observational
Sponsor: The Lymphoma Academic Research Organisation (Other)
Responsible Party: Sponsor
Other Study IDs: ADAMANTIUS
Record Dates: First submitted 2014-09-11; First posted 2014-11-25 (Estimated); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Hodgkin Lymphoma; B-Cell Lymphoma
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, B-Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The present study aims to further optimize a whole-body Diffusion-Weighted Magnetic Resonance Imagery (DW-MRI or DWI) protocol on 3 Tesla MR and/or new system combining 3Tesla MR and Positron Emission Tomography (PET), to develop and validate an automated whole-body parametric image analysis algorithm, and to determine the added value of whole-body DWI to Fluorodeoxyglucose-PET for the management of lymphoma patients.

DETAILED DESCRIPTION:
Imaging biomarkers are important tools for the detection and characterization of cancers as well as for monitoring the response to therapy. "Whole-body" molecular imaging, in particular using 18-Fluorodeoxyglucose-PET, has been proven useful in the evaluation and management of lymphoma patients. FDG-PET has evolved as a valuable biomarker in aggressive lymphomas, which is the current state-of-the-art imaging technique for response assessment at the end of treatment. Additionally, the prognostic value of "interim" (during treatment) or early PET has been well established in Hodgkin lymphoma and diffuse large B-cell lymphoma, which together account for more than 50% of all lymphomas. Worldwide clinical trials are ongoing to evaluate risk-adapted individualized treatment strategy based on interim PET results. Therefore, uniform and evidence-based guidelines for the interpretation are warranted. International Workshop on Interim PET in Lymphoma recently proposed a 5-point score method and so far the results of validation studies are promising.

However, one could speculate that the risk of false-positive studies due to a non-specific inflammatory effect will be greater when patients receiving more toxic regimens and the usefulness of imaging biomarkers would vary for different lymphoma subtypes. Meanwhile, thanks to rapid technical development, whole-body functional magnetic resonance imaging (MRI) in particular diffusion-weighted MRI (DWI) reflecting cell density is now feasible in the clinical setting. Quantitative parameters derived from DWI reflecting cell density may provide complementary information to current state-of-the-art FDG-PET imaging reflecting quantitatively glucose metabolism and prove to be helpful in patient management.

Pilot studies have shown the potential of whole-body DWI in lymphomas for staging and response assessment on 1.5 Tesla MR system but larger-scaled prospective studies are required before this new imaging-based biomarker can ever be validated for routine clinical use. Besides, technical challenges remain especially when encountering higher-field clinical MR systems. Finally, a vast amount of information generated from whole-body parametric imaging data will require development of automated image analysis software, which may help in establishing a multi-parametric approach in characterizing residual lymphoma masses.

Therefore, the present study aims to further optimize a whole-body DWI protocol on 3 Tesla MR and/or new system combining 3Tesla MR and PET, to develop and validate an automated whole-body parametric image analysis algorithm, and to determine the added value of whole-body DWI to FDG-PET for the management of lymphoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed hodgkin's lymphoma, diffuse large B-cell lymphoma or follicular lymphoma
* Patients aged over 18
* Initial presentation of bulky disease

Exclusion Criteria:

* Patients with impaired central nervous system
* Patients regularly taking corticosteroids during the 4 weeks preceding the treatment (unless the dose administered is equivalent to ≤20 mg/day prednisone).
* Patients who have undergone major surgery during the 28 days preceding the inclusion
* Patients with low kidney and/or liver function
* Patients with HIV +
* Patients whose life expectancy ≤ 6 months
* Patients with other medical problems or psychological susceptibles interfere with the study,
* Patients under adult supervision.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed HL, DLBCL or FL At least 18 years of age Initial presentation of bulky disease
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2014-10; Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
apparent diffusion coefficient changes of post-treatment residual lymphoma masses and whether this MR-derived parameter helps in characterizing its viability in addition to PET | Baseline
correlation between standardized uptake value and apparent diffusion coefficient changes; correlation with post-treatment histopathological findings if tissue proof | Baseline, 6 weeks, between 18 and 24 weeks
correlation between the PET and MR-derived functional parameters with clinical outcome (end-treatment response and survival) | Between 18 and 24 weeks

OTHER OUTCOMES:
development of automated lesion detection algorithm | Baseline, 6 weeks, between 18 and 24 weeks
texture analysis of the major lymphoma mass and correlation of tumor heterogeneity with treatment outcome | Baseline, 6 weeks, between 18 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alain Rahmouni, Prof., Principal Investigator — CHU Henri Mondor; Corinne Haioun, Prof., Principal Investigator — Lymphoma Study Association; Emmanuel Itti, Prof., Principal Investigator — CHU Henri Mondor
Locations (1):
- Hopital Henri Mondor, Créteil, France

IPD SHARING:
Plan to Share IPD: No